CLINICAL TRIAL: NCT03564834
Title: Laparoscopic Versus Open Gastrectomy for Elderly Local Advanced Gastric Cancer Patients: a Phase II Randomized Parallel Controlled Trial
Brief Title: Laparoscopic Versus Open Gastrectomy for Elderly Local Advanced Gastric Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, Deputy Director of Department of Surgery, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF2018-4-2156
Record Dates: First submitted 2018-05-14; First posted 2018-06-21 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Advanced Gastric Cancer
Keywords: Elderly patients; Open gastrectomy; Laparoscopic gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic gastrectomy (Experimental): A standard laparoscopic gastrectomy with D2 lymphadenectomy will be performed by two experienced surgeons, according to the Japanese Gastric Cancer Treatment Guidelines 2014 (version 4) and the Japanese Classification of Gastric Carcinoma (3rd English edition).
  Interventions: Procedure: Laparoscopic gastrectomy
- Open gastrectomy (Active Comparator): A standard open gastrectomy with D2 lymphadenectomy will be performed by two experienced surgeons, according to the Japanese Gastric Cancer Treatment Guidelines 2014 (version 4) and the Japanese Classification of Gastric Carcinoma (3rd English edition).
  Interventions: Procedure: Open gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — Patients will receive laparoscopic gastrectomy within one week after randomization.
  Arms: Laparoscopic gastrectomy
Procedure: Open gastrectomy — Patients will receive open gastrectomy within one week after randomization.
  Arms: Open gastrectomy

SUMMARY:
Gastric cancer is one of the most common malignant tumors worldwide. With the rapid aging of global population, the number of elderly patients with local advanced gastric cancer is increasing. Surgery is the essential treatment for local advanced gastric cancer. However, because of the degeneration of physiological organs, cell functions, compensatory ability, immunity, and physiological reserve ability, elderly patients often face great safety issues when having surgery. Therefore, how to treat the elderly patients with local advanced gastric cancer with safe and effective surgery is one of the important problems in the field of gastric cancer treatment. With the introduction of minimally invasive treatment concepts and techniques, the role of laparoscopic radical gastrectomy in the treatment of early gastric cancer, as well as the advantages of trauma control and postoperative accelerated rehabilitation have been confirmed, however, there is still a lack of sufficient high-level clinical evidence in the elderly patients with advanced gastric cancer. The current study therefore aims to evaluate the safety and efficacy of laparoscopic versus open gastrectomy for advanced gastric cancer in elderly patients, using a randomized parallel controlled study design. The investigators hypothesized that laparoscopic gastrectomy is superior to open gastrectomy in terms of perioperative safety for local advanced gastric cancer patients aged 70 and above.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common cancer and cause of cancer death worldwide. With the rapid aging of global population, the number of elderly patients with local advanced gastric cancer has been continuously increasing. Surgery is the essential treatment for local advanced gastric cancer. However, elderly patients are at high risk of postoperative complications due to reduced functional reserve and increased comorbidities. Studies have shown that elder patients can have postoperative complication incidence up to 18%-32% and surgery-related mortality rate to 3.8%-9.5%. Therefore, elderly patients usually require more restrict operative injury control compared to the younger population. Surgical safety and effectiveness has become a crucial research focus for local advanced gastric cancer among elderly patients.

Laparoscopic gastrectomy is one of the standard treatments for early gastric cancer and has demonstrated its application value in local advanced gastric cancer. Two recent meta-analysis on observational studies have shown the feasibility of laparoscopic gastrectomy in elderly gastric cancer patients. Compared to conventional open resections, elderly patients may benefit from the advantages of laparoscopic approach such as less trauma, less blood loss, faster bowel movement recovery, earlier food intake, and shorter hospitalization. However, laparoscopic gastrectomy raises issues such as prolonged operation time and disturbance of circulatory and respiratory dynamics by carbon dioxide pneumoperitoneum during the procedure. Nonetheless, all currently available evidence comes from observational studies that are susceptible to bias and evidence on long-term survival is scarce. The investigators therefore proposed to conduct this randomized controlled trial comparing the feasibility and survival benefit of laparoscopic with open gastrectomy for elderly patients with local advanced gastric cancer. The investigators hypothesized that laparoscopic gastrectomy is superior to open gastrectomy in terms of perioperative safety for local advanced gastric cancer patients aged 70 and above.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female aged 70 and above
* Karnofsky score≥70%
* Histologically proven gastric adenocarcinoma in biopsy (including Lauren classification) Proven clinical stage of cT2-4aNanyM0 by baseline ultrasound endoscope, enhanced CT/MRI examination, or diagnostic laparoscopy using Habermann Standards
* No past chemotherapy or radiotherapy before diagnosis
* Primary tumor located at stomach, achievable naked-eye complete resection (R0/1) via distal subtotal or total gastrectomy plus lymphadenectomy
* Haematology and biochemistry index meet the following: hemoglobin≥80g/L, absolute neutrophils count (ANC)≥1.5×109/L, platelet≥100×109/L, ALT、AST≤2.5 times the upper limit of normal value, ALP≤2.5 times the upper limit of normal value, serum total bilirubin<1.5 times the upper limit of normal value, serum creatinine<1 times the upper limit of normal value, serum albumin≥30g/L
* Heart and lung function can withstand surgery
* No severe concomitant disease that leads to survival<3 years
* Willing and able to comply with study protocol Written agreement consent before enrolment and full aware of the right to quit the study at any time with no loss

Exclusion Criteria:

* Uncontrolled seizure, central nervous system diseases, or mental disorders;
* Past history of upper abdominal surgery (except for laparoscopic cholecystectomy)
* Past history of gastric surgery (including diagnosis procedure such as ESD and EMR)
* Other malignant diseases in 5 years (except for cured skin carcinoma and cervical carcinoma in situ)
* Clinical severe or active heart diseases, such as symptomatic coronary heart disease, NYHA grade II or above congestive heart failure, severe arrhythmia, or myocardial infarction in 6 months
* Cerebral hemorrhage or infarction in 6 months
* Organ transplant recipients under immunosuppressive therapy
* Severe uncontrolled repeated infection or other severe uncontrolled concomitant diseases
* Medium or severe renal damage (creatinine clearance rate≤50ml/min or serum creatinine> upper limit of normal value)
* Other diseases requiring synchronous surgery
* Requiring emergent surgery due to oncologic emergent (e.g. bleeding, perforation, obstruction)
* FEV1<50% of expected value Participated in other studies 4 weeks before the randomization.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rate | within 30 days after surgery
  Surgery related complications include incision complications (infection, effusion, dehiscence, poor healing), peritoneal effusion or abscess formation, hemorrhage (inside abdominal cavity, inside digestive tract), ileus, anastomotic leakage, anastomotic stenosis, intestinal fistula, lymphatic leakage, pancreatic fistula, gastroparesis, pancreatitis, lung infection, pleural effusion, urinary tract infection, renal failure, liver failure, cardio-cerebrovascular events (both lower extremities thrombosis, pulmonary embolism, myocardial infarction, arrhythmia, cerebral infarction, etc.), and others. Complications will be reported and graded according to the Clavien-Dindo classification of surgical complications.

SECONDARY OUTCOMES:
Length of postoperative hospitalization stay | within 30 days after surgery
  Postoperative hospitalization stay refers to the time interval between the day of surgery and discharge, and will be recorded by the investigators.
Postoperative life quality | one-year after surgery
  Will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaires (i.e. QLQ-C30), which contains both QLQ-STO22 and ELD14 modules. This is a questionnaire developed to assess the generic and disease-specific quality of life for elderly gastric cancer patients by European Organisation for Research and Treatment of Cancer. The Summary Score will be calculated from the mean of scales. Prior to calculating the mean, the symptom scales will need to be reversed to obtain a uniform direction of all scales. The summary score should only be calculated if all of the required scale scores are available (using scale scores based on the completed items, provided that at least 50% of the items in that scale have been completed.
Three-year overall survival rate | Three-year after surgery
  Overall survival is defined as the time interval from the time of the radical gastrectomy to the date of all-cause death or the last follow-up. Three-year overall survival rate will be calculated using the Kaplan-Meier Methods.
Three-year disease-free survival rate | Three-year after surgery
  Disease-free survival is defined as the time interval from the time of the radical gastrectomy to the date of the detection of cancer recurrence or the last follow-up. Three-year disease-free survival rate will be calculated using the Kaplan-Meier Methods.
Postoperative pain | within 2 weeks after surgery
  Postoperative pain will be measured using the Numeric Rating Scale (NRS-11) which is an 11-point scale for patient self-reporting of pain. The scale ranges from 0 to 10, with 0 being no pain. Pain level will be graded into four levels for analysis: "0: No Pain", "1-3: Mild Pain", "4-6 Moderate Pain", and "7-10 Severe Pain".

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, MD, Principal Investigator — Peking University Cancer Hospital and Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The deidentified datasets generated during the current study will be publicly available via an appropriate data archive 6 months after the completion of the trial.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after the completion of the trial
Access Criteria: As request

REFERENCES:
- [Derived] Li Z, Shan F, Ying X, Xue K, Ji J. Laparoscopic versus open gastrectomy for elderly local advanced gastric cancer patients: study protocol of a phase II randomized controlled trial. BMC Cancer. 2018 Nov 16;18(1):1118. doi: 10.1186/s12885-018-5041-y. PMID 30445943